CLINICAL TRIAL: NCT05631756
Title: "Correlation Between PaO2/FiO2 and Lung Ultrasound Score in Patients Admitted to an Intensive Care Unit With Interstitial Syndrome: A Prospective Physiological Study"
Brief Title: Correlation Between PaO2/FiO2 and Lung Ultrasound Score in the Intensive Care Unit
Acronym: O2LUSSU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022/24NOV/444
Record Dates: First submitted 2022-10-13; First posted 2022-11-30 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Population (Experimental): All patients included in the study, meaning patients in the ICU presenting an interstitial syndrom no matter the aetiology
  Interventions: Other: Lung Ultrasound

INTERVENTIONS:
Other: Lung Ultrasound — Evaluation of the Lung Ultrasound Score in patients presenting an interstitial syndrom on the lung ultrasound and to compare it with PaO2/FiO2

SUMMARY:
The goal of this physiological interventional prospective study is to evaluate the improvement of the previously demonstrated correlation between PaO2/ FiO2 and Lung Ultrasound score (LUSS) in patients admitted in the ICU with an intesrtitial syndrom (IS) on the ultrasound of all aetiologies at inclusion and at twenty four and forty eight hours.

The main question it aims to answer is if the LUSS is a valid tool to evaluate the severity of the IS Participants will initially have an arterial blood gas to evaluate the PaO2/FiO2 and in the ten minutes a lung ultrasound to evaluate the LUSS. This will be repeated at twenty four and forty eight hours.

DETAILED DESCRIPTION:
JUSTIFICATION FOR THE RESEARCH

Interstitial Syndrome (IS) also known as alveolar-interstitial syndrome, is a diffuse affection of the lung interstitial tissue leading to decreased alveolo-capillary exchange and therefore hypoxemia. Acute conditions such as viral or bacterial pneumonia and pulmonary edema lead to IS. Pulmonary edema can either be haemodynamically induced in acute heart failure (AHF) or secondary to permeability impairment in Acute Respiratory Distress Syndrome (ARDS). In literature, Acute Lung Injury (ALI) is also used to refer to a condition similar to ARDS with less severe hypoxemia. Chronic pathologies as Diffuse Parenchymal Lung Disease (DPLD) also cause IS. Lung Ultrasound (LUS) is a useful tool to diagnose IS. Indeed, LUS is non-invasive, non-irradiating, low cost and easily available at the patient's bedside. The interest of LUS for critically ill patient has been demonstrated5. In ICU, it was shown that LUS reduces number of chest radiography, relative medical costs and radiation exposure without affecting patient outcome. Literature suggests that LUS diagnostic accuracy for IS is higher than the diagnostic accuracy of chest radiography. Chest Computed Tomography is the actual gold standard for IS diagnosis, however not available at patient bedside, irradiating and more expensive. LUS is mostly based on the detection of artefacts created by air-tissue interfaces5. In IS, artefacts have been shown to be related to the presence of extra-vascular water and the water-thickened of interlobular septa. Comet Tail Artefact (CTA) was originally described as dense tapering trail of echoes just distal to a strongly reflective surface whereas Ring Down Artefact (RDA) starts from the point of origin of the ultrasound waves and "ring-down" to the end of the screen without fading. CTA and RDA are created by different mechanisms. Liechtenstein's early work introduced the term CTA to describe artefacts found in IS4. He later introduced the alphabetic nomenclature and assign the term B-lines to those IS artefacts. According to Yue Lee and All, a confusion between CTA and RDA exist in the literature as B-Lines definition correspond to RDA rater then CTA. International recommendations later agreed on the use of the term B-line, to describe artefact found in IS. Presence of multiple B-lines is widely recognised to suggest the presence of IS. Despite poor literature on this topic, IS severity is represented by hypoxemia generally evaluated by the realization of an Arterial Blood Gase (ABG) to obtain Arterial Partial Pressure in Oxygen (PaO2). A study however supported the absence of correlation between PaO2 and long-term mortality for AHF. Another rather recent study, including one-hundred and sixty-five COVID-19 patients that underwent non-invasive ventilation, nevertheless showed a statistically significant difference in PaO2 between survivor and non-survivor at twenty-eight days. According to the Berlin definition, hypoxemia represented by the ratio between PaO2 and the fraction of inspired oxygen (FiO2) is a severity indicator in ARDS. LUS could be an alternative to evaluate severity of IS. The Lung Ultrasound Score (LUSS) was initially developed on an experimental model to assess lung aeration and is based on quantitative assessment of B-lines in six thoracic zones bilaterally. In each zone, a sonographic lung aeration status is determined scoring from zero to four to determine a total score over thirty-six. Literature findings are consistent with LUSS being an efficient tool to measure lung aeration in different intensive care situations: re-aeration antibiotics-induced in Ventilator Associated Pneumonia, assessment of PEEP-induced lung recruitment. LUSS realized during weaning trial has been showed to be able to predict of postextubation distress. In the Intensive Care Unit (ICU), LUSS is efficient to quantify lesions and predict mortality associated with ARDS. During the recent COVID-19 pandemic, numerous trials have demonstrated that LUSS is associated with disease severity and mortality in COVID-19 patients. Recently, a negative linear correlation between PaO2/FiO2 and LUSS was shown three series of patients admitted to Intensive Care Units (ICU) with different aetiologies of IS: one with thirty-three COVID-19 patients, one with thirty-seven ARDS patients and one with seventy-two ALI patients. Lately, this correlation was confirmed in larger series of one-hundred and sixty-two patients admitted the Emergency Departement (ED) suggesting that LUSS could be a tool to evaluate PaO2 and therefore evaluate IS severity regardless of IS' aetiology in patients admitted to ED.

STUDY PROCEDURE

A LUSS will be realized by an investigator trained for Lung UltraSound (LUS) and considering him/herself confident for its use. A five-point Likert scale will be filled. To the statement "I am qualified to realize a LUSS", only emergency doctors answering "I strongly agree" or "I agree" will be eligible for inclusion and added to investigators list using an amendment to this protocol. The ultrasound machines operated for LUS belong to each ED meaning the investigators are familiar to its use. To uniformize the results, settings of the ultrasound machines will be standardized. To allow the exploration of the pulmonary parenchyma a low frequency curvilinear transducer will be used, and evaluation of B-lines will be performed using a depth of at least 12cm as commonly recommended. If patients are isolated for infectious reasons, special precautions will be applied following institutional procedures of ultrasound use on contagious patients. LUS will take place within 10 minutes of ABG analysis. LUS will be performed at the patient's bedside. The investigator will be blinded to any other procedure made by treating physician for diagnostic purposes. The treating physician will be allowed to perform a LUS on its own. The LUSS procedure will be used as validated in a larger number of studies. For that matter, the thorax is virtually divided in six thoracic zones bilaterally, comporting two anterior zones, two lateral zones and two posterior zones. The anterior and lateral zones will be evaluated in strict dorsal decubitus and the posterior zones will be evaluated with a light contro-lateral decubitus allowed, if necessary, because of patient morphotype.

For each zone a score from zero to three will be determined as shown in figure 4:

* 0: A normal aeration of the lung with presence of A lines, persistent pleural sliding and less than three B-lines.
* 1: Interstitial syndrome, resulting in moderate loss of aeration with more than three spaced B-lines, 7mm apart, scores one point.
* 2: Alveolar-interstitial syndrome meaning a severe loss of aeration with coalescent B-lines, less then 3mm apart, scores two.
* 3: An alveolar consolidation leading to a complete loss of aeration with an ultrasonographic tissue like pattern.

LUSS will be calculated by adding the score given to each 12 zones, with a maximum of thirty-six. Patients scoring less than two, will be considered empirically with no interstitial syndrome and will be excluded of the study.

Investigators will also report the presence of pleural effusions and if present estimate their amount. If present, pleural effusions quantification will be realized at lung base. The maximal distance between parietal and visceral pleura (Dmax) in millimeter will be measured after freezing the image in end-expiration.

If the ABG indication according to treating ICU physician persist, the complete intervention including calculation of LUSS, research and quantification of pleural effusions will be repeated at twenty-four and forty-eight hours.

Result of LUSS, pleural effusions' presence and Dmax won't be communicated to the treating physician expect if the LUS results could influence patient prognosis.

STUDY CONDUCTION

Study Settings:

Before the study launching, the investigator will be evaluated using a five-point Likert scale as previously described. A presentation of the study and the procedure will be organized by the coordinating investigators in each center.

Patients' recruitment:

The eligible patients will be identified by the treating ICU physician. Adult patients admitted to ICU with signs and symptoms of ARF and an indication of realization of ABG to evaluate PaO2 according to treating ICU physician will be considered for inclusion. ABG won't be considered as an intervention as the decision of the realization of an ABG is being left to the treating ICU physician. If those criteria are met, treating physician will contact an investigator.

Inclusion:

Investigator will be responsible to verify if patient meet all inclusion criteria. Consent will correspond to the signature of a paper consent form in duplicate after being informed over research modalities by the investigator. If the patient is unable to give his consent because of an acute condition and have no legal representative, a delayed consent will be authorized. One signed copy of the consent form will be returned to the patient or the legal representative.

Intervention:

All included patients will undergo a LUS, the calculation of a LUSS and search of pleural effusions and pleural effusions' quantification by Dmax measurement when pleural effusions are present. In Belgium, LUS isn't recognized as standard of care giving to this study an interventional character. Intervention will take place in a range of time of maximum then minutes before or after ABG realization. The result of the intervention will not be communicated to the treating physician except when LUS could influence patient's prognosis.

Follow up:

If ABG indication persists following treating ICU physician and if the patient is still present in the ICU, the intervention as described previously will be repeated at twenty-four and forty-eight hours.

Data collection and Data treatment:

After inclusion data will be reported in an informatized CRF using REDCap software by investigator and Pleural Effusion Volume (Vpe) in milliliter will be automatically calculated by multiplying Dmax per twenty according to Balik and all's formula. The SOFA score at inclusion, twenty-four and forty-eight hours will also be calculated and recorded. Name, first name, date of birth and hospital administrative number of the included patients will be recorded. Investigators will only access personal data of the patient they have personally included. Principal investigators will have access to all personal data to be able to collect missing data. After data completion, a neutral identifier composed by inclusion centre's number, number of inclusion and year of birth will be used. A correspondence list will be kept under the principal investigator responsibility.

STATISTICS

Data analysis was performed using JMP Pro 16.0.0 Software (SAS Institute). Continuous variables are expressed as mean values and standard deviations. Discrete variables are reported as categories and expressed as numbers and percentages. The Pearson correlation was used to measure the linear correlation between continuous variables, and correlations are expressed as correlation coefficient and 95% confidence interval. Comparisons between quantitative data were performed with a χ2 test, and between-group comparisons between continuous data with a Wilcoxon-Mann-Whitney test. The significance threshold was set with a P value of < 0.05. A one-sided hypothesis test will be use to show the improvement of the correlation between PaO2/FiO2 and LUSS. Pearson formula will be used to show correlation between PaO2/FiO2 and LUSS. Multiple linear regression will be used to test the effects of continuous variables such as presence of pleural effusions on the correlation between PaO2/FIO2 and LUSS.

ELIGIBILITY:
Inclusion Criteria:

- consent

->17 years old

Exclusion Criteria:

* LUSS < 2

Non Inclusion Criteria:

* Patient with pathologies leading to chronic IS
* Chronic Obstructive Pulmonary Disease (COPD) or active asthma
* Patients under veino-veinous or veino-arterial " Extracorporeal Membrane Oxygenation " (ECMO)
* Severe trauma patients
* Less than twenty-four hours post operative patients
* LUS not feasible: prone position, pneumonectomy history, severe obesity

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Correlation PaO2/FiO2 and LUSS | At inclusion
  To assess the correlation between the PaO2/FiO2 and the LUSS in patients admitted in an ICU with IS.

SECONDARY OUTCOMES:
Evolution | Twenty four and forty eight hours
  To assess the evolution of the correlation between the PaO2/FiO2 and the LUSS at inclusion, twenty-four hours, and forty-eight hours after inclusion in patients admitted in an ICU with IS.
Lung Ultrasound Score and SOFA score | Inclusion,twenty four and forty eight hours
  to assess the presence of a correlation between LUSS and the SOFA score at inclusion, twenty-four et forty-eight hours of inclusion in patient admitted to an ICU with IS.
Influence SOFA on the correlation between PaO2/FiO2 and LUSS | Inclusion,twenty four and forty eight hours
  To determine the influence of the SOFA score on the correlation between PaO2/FiO2 and LUSS at inclusion, twenty-four et forty-eight hours of inclusion in patients admitted to an ICU with IS.
Pleural Effusions | Inclusion, twenty four and forty eight hours
  To to determine the influence of the presence and size of pleural effusions on the correlation between PaO2/FiO2 and LUSS at inclusion, twenty-four et forty-eight hours of inclusion in patients admitted to an ICU with IS.
Correlation PaO2/FiO2 and the LUSS according to IS diagnosis | Inclusion
  To assess the correlation between the PaO2/FiO2 and the LUSS in patients admitted in an ICU with IS According to the aetiologic diagnosis attributed to the IS (pulmonary oedema, bacterial or viral infection, post operative reactionary hypoventilation)
  The end point of this secondary outcome considers the null hypothesis to be an improvement of 0,214 of the correlation between PaO2/FiO2 and LUSS
Correlation between the PaO2/FiO2 and the LUSS admission diagnosis | Inclusion
  To assess the correlation between the PaO2/FiO2 and the LUSS in patients admitted in an ICU with IS according to admission diagnosis (cardiogenic shock, sepsis, infection, post operative)
Correlation between the PaO2/FiO2 and the LUSS according to the LUSS value | Inclusion
  To assess the correlation between the PaO2/FiO2 and the LUSS in patients admitted in an ICU with IS according to LUSS value (between two and six and between seven and thirty-six) The end point of this secondary outcome considers a negative linear distribution for PaO2/FiO2 and LUSS values
Correlation between the PaO2/FiO2 and LUSS according to hypoxemia | Inclusion
  To assess the correlation between the PaO2/FiO2 and the LUSS in patients admitted in an ICU with IS acordiing on hypoxemia severity based on PaO2/FiO2 as defined for ARDS3 (mild hypoxemia with PaO2/FiO2 between three hundred and two hundred, moderate hypoxemia with PaO2/FiO2 between one hundred and two hundred and severe hypoxemia with a PaO2/FiO2 of less than one hundred)
Correlation between the PaO2/FiO2 and LUSS according to the RR at admission | Inclusion
  To assess the correlation between the PaO2/FiO2 and the LUSS in patients admitted in an ICU with IS according to Respiratory Rate (RR) (low RR of less than twelve per minute, normal RR between twelve and twenty and elevated RR of more than twenty)
Evolution of the correlation between the PaO2/FiO2 and the LUSS according to IS diagnosis | Twenty four and forty eight hours
  To assess the evolution of the correlation between the PaO2/FiO2 and the LUSS at inclusion, twenty-four hours, and forty-eight hours after inclusion in patients admitted in an ICU with IS According to the aetiologic diagnosis attributed to the IS (pulmonary oedema, bacterial or viral infection, post operative reactionary hypoventilation) a negative linear distribution for PaO2/FiO2 and LUSS values
Evolution of the correlation between the PaO2/FiO2 and the LUSS according to admission diagnosis | Twenty four and forty eight hours
  To assess the evolution of the correlation between the PaO2/FiO2 and the LUSS at inclusion, twenty-four hours, and forty-eight hours after inclusion in patients admitted in an ICU with IS according to admission diagnosis (cardiogenic shock, sepsis, infection, post operative)
Evolution of the correlation between the PaO2/FiO2 and the LUSS according to LUSS value | Twenty four and forty eight hours
  To assess the evolution of the correlation between the PaO2/FiO2 and the LUSS at inclusion, twenty-four hours, and forty-eight hours after inclusion in patients admitted in an ICU with IS according to LUSS value (between two and six and between seven and thirty-six)
Evolution of the correlation between the PaO2/FiO2 and the LUSS according to hypoxemia severity | Twenty four and forty eight hours
  To assess the evolution of the correlation between the PaO2/FiO2 and the LUSS at inclusion, twenty-four hours, and forty-eight hours after inclusion in patients admitted in an ICU with IS acordiing on hypoxemia severity based on PaO2/FiO2 as defined for ARDS3 (mild hypoxemia with PaO2/FiO2 between three hundred and two hundred, moderate hypoxemia with PaO2/FiO2 between one hundred and two hundred and severe hypoxemia with a PaO2/FiO2 of less than one hundred)
Evolution of the correlation between the PaO2/FiO2 and the LUSS according RR | Twenty four and forty eight hours
  To assess the evolution of the correlation between the PaO2/FiO2 and the LUSS at inclusion, twenty-four hours, and forty-eight hours after inclusion in patients admitted in an ICU with IS according to Respiratory Rate (RR) (low RR of less than twelve per minute, normal RR between twelve and twenty and elevated RR of more than twenty)
Correlation between LUSS and the SOFA score at inclusion according to the diagnosis of the IS | Inclusion,twenty four and forty eight hours
  To assess the presence of a correlation between LUSS and the SOFA score at inclusion, twenty-four et forty-eight hours of inclusion in patient admitted to an ICU with IS According to the aetiologic diagnosis attributed to the IS (pulmonary oedema, bacterial or viral infection, post operative reactionary hypoventilation) The end point of this secondary outcome considers a positive linear correlation between LUSS and SOFA score and a negative linear distribution for the correlation between PaO2/FiO2 and LUSS corrected by the SOFA score
Correlation between LUSS and the SOFA score at inclusion according to admission diagnosis | Inclusion,twenty four and forty eight hours
  to assess the presence of a correlation between LUSS and the SOFA score at inclusion, twenty-four et forty-eight hours of inclusion in patient admitted to an ICU with IS according to admission diagnosis (cardiogenic shock, sepsis, infection, post operative) The end point of this secondary outcome considers a positive linear correlation between LUSS and SOFA score and a negative linear distribution for the correlation between PaO2/FiO2 and LUSS corrected by the SOFA score
Correlation between LUSS and the SOFA score according to the LUSS value | Inclusion,twenty four and forty eight hours
  to assess the presence of a correlation between LUSS and the SOFA score at inclusion, twenty-four et forty-eight hours of inclusion in patient admitted to an ICU with IS according to LUSS value (between two and six and between seven and thirty-six) The end point of this secondary outcome considers a positive linear correlation between LUSS and SOFA score and a negative linear distribution for the correlation between PaO2/FiO2 and LUSS corrected by the SOFA score
Correlation between LUSS and the SOFA score according to hypoxemia severity | Inclusion,twenty four and forty eight hours
  to assess the presence of a correlation between LUSS and the SOFA score at inclusion, twenty-four et forty-eight hours of inclusion in patient admitted to an ICU with IS acordiing on hypoxemia severity based on PaO2/FiO2 as defined for ARDS3 (mild hypoxemia with PaO2/FiO2 between three hundred and two hundred, moderate hypoxemia with PaO2/FiO2 between one hundred and two hundred and severe hypoxemia with a PaO2/FiO2 of less than one hundred) The end point of this secondary outcome considers a positive linear correlation between LUSS and SOFA score and a negative linear distribution for the correlation between PaO2/FiO2 and LUSS corrected by the SOFA score
Correlation between LUSS and the SOFA score according to the RR | Inclusion,twenty four and forty eight hours
  to assess the presence of a correlation between LUSS and the SOFA score at inclusion, twenty-four et forty-eight hours of inclusion in patient admitted to an ICU with IS according to Respiratory Rate (RR) (low RR of less than twelve per minute, normal RR between twelve and twenty and elevated RR of more than twenty) The end point of this secondary outcome considers a positive linear correlation between LUSS and SOFA score and a negative linear distribution for the correlation between PaO2/FiO2 and LUSS corrected by the SOFA score
Influence of the SOFA score on the correlation between PaO2/FiO2 and LUSS according to IS diagnosis | Inclusion,twenty four and forty eight hours
  To determine the influence of the SOFA score on the correlation between PaO2/FiO2 and LUSS at inclusion, twenty-four et forty-eight hours of inclusion in patients admitted to an ICU with IS According to the aetiologic diagnosis attributed to the IS (pulmonary oedema, bacterial or viral infection, post operative reactionary hypoventilation) The end point of this secondary outcome considers a positive linear correlation between LUSS and SOFA score and a negative linear distribution for the correlation between PaO2/FiO2 and LUSS corrected by the SOFA score
Influence of the SOFA score on the correlation between PaO2/FiO2 and LUSS according to admission diagnosis | Inclusion,twenty four and forty eight hours
  To determine the influence of the SOFA score on the correlation between PaO2/FiO2 and LUSS at inclusion, twenty-four et forty-eight hours of inclusion in patients admitted to an ICU with ISaccording to admission diagnosis (cardiogenic shock, sepsis, infection, post operative) The end point of this secondary outcome considers a positive linear correlation between LUSS and SOFA score and a negative linear distribution for the correlation between PaO2/FiO2 and LUSS corrected by the SOFA score
Influence of the SOFA score on the correlation between PaO2/FiO2 and LUSS according to LUSS value | Inclusion,twenty four and forty eight hours
  To determine the influence of the SOFA score on the correlation between PaO2/FiO2 and LUSS at inclusion, twenty-four et forty-eight hours of inclusion in patients admitted to an ICU with IS according to LUSS value (between two and six and between seven and thirty-six) The end point of this secondary outcome considers a positive linear correlation between LUSS and SOFA score and a negative linear distribution for the correlation between PaO2/FiO2 and LUSS corrected by the SOFA score
Influence of the SOFA score on the correlation between PaO2/FiO2 and LUSS according to hypoxemia severity | Inclusion,twenty four and forty eight hours
  To determine the influence of the SOFA score on the correlation between PaO2/FiO2 and LUSS at inclusion, twenty-four et forty-eight hours of inclusion in patients admitted to an ICU with IS acordiing on hypoxemia severity based on PaO2/FiO2 as defined for ARDS3 (mild hypoxemia with PaO2/FiO2 between three hundred and two hundred, moderate hypoxemia with PaO2/FiO2 between one hundred and two hundred and severe hypoxemia with a PaO2/FiO2 of less than one hundred) The end point of this secondary outcome considers a positive linear correlation between LUSS and SOFA score and a negative linear distribution for the correlation between PaO2/FiO2 and LUSS corrected by the SOFA score
Influence of the SOFA score on the correlation between PaO2/FiO2 and LUSS according to RR | Inclusion,twenty four and forty eight hours
  To determine the influence of the SOFA score on the correlation between PaO2/FiO2 and LUSS at inclusion, twenty-four et forty-eight hours of inclusion in patients admitted to an ICU with IS.according to Respiratory Rate (RR) (low RR of less than twelve per minute, normal RR between twelve and twenty and elevated RR of more than twenty) The end point of this secondary outcome considers a positive linear correlation between LUSS and SOFA score and a negative linear distribution for the correlation between PaO2/FiO2 and LUSS corrected by the SOFA score
Influence of the presence and size of pleural effusions on the correlation between PaO2/FiO2 and LUSS according to IS diagnosis | Inclusion,twenty four and forty eight hours
  To determine the influence of the presence and size of pleural effusions on the correlation between PaO2/FiO2 and LUSS at inclusion, twenty-four et forty-eight hours of inclusion in patients admitted to an ICU with IS According to the aetiologic diagnosis attributed to the IS (pulmonary oedema, bacterial or viral infection, post operative reactionary hypoventilation) The end point of this secondary outcome considers a negative linear distribution for the correlation between PaO2/FiO2 and LUSS corrected by the presence of pleural effusions and pleural effusions' size.
Influence of the presence and size of pleural effusions on the correlation between PaO2/FiO2 and LUSS according to admission diagnosis | Inclusion,twenty four and forty eight hours
  To determine the influence of the presence and size of pleural effusions on the correlation between PaO2/FiO2 and LUSS at inclusion, twenty-four et forty-eight hours of inclusion in patients admitted to an ICU with IS according to admission diagnosis (cardiogenic shock, sepsis, infection, post operative) The end point of this secondary outcome considers a negative linear distribution for the correlation between PaO2/FiO2 and LUSS corrected by the presence of pleural effusions and pleural effusions' size.
Influence of the presence and size of pleural effusions on the correlation between PaO2/FiO2 and LUSS according to LUSS value | Inclusion,twenty four and forty eight hours
  To determine the influence of the presence and size of pleural effusions on the correlation between PaO2/FiO2 and LUSS at inclusion, twenty-four et forty-eight hours of inclusion in patients admitted to an ICU with IS according to LUSS value (between two and six and between seven and thirty-six) The end point of this secondary outcome considers a negative linear distribution for the correlation between PaO2/FiO2 and LUSS corrected by the presence of pleural effusions and pleural effusions' size.
Influence of the presence and size of pleural effusions on the correlation between PaO2/FiO2 and LUSS according to hypoxemia severity | Inclusion,twenty four and forty eight hours
  To determine the influence of the presence and size of pleural effusions on the correlation between PaO2/FiO2 and LUSS at inclusion, twenty-four et forty-eight hours of inclusion in patients admitted to an ICU with IS acordiing to hypoxemia severity based on PaO2/FiO2 as defined for ARDS3 (mild hypoxemia with PaO2/FiO2 between three hundred and two hundred, moderate hypoxemia with PaO2/FiO2 between one hundred and two hundred and severe hypoxemia with a PaO2/FiO2 of less than one hundred) The end point of this secondary outcome considers a negative linear distribution for the correlation between PaO2/FiO2 and LUSS corrected by the presence of pleural effusions and pleural effusions' size.
Influence of the presence and size of pleural effusions on the correlation between PaO2/FiO2 and LUSS according to RR | Inclusion,twenty four and forty eight hours
  To the influence of the presence and size of pleural effusions on the correlation between PaO2/FiO2 and LUSS at inclusion, twenty-four et forty-eight hours of inclusion in patients admitted to an ICU with IS according to Respiratory Rate (RR) (low RR of less than twelve per minute, normal RR between twelve and twenty and elevated RR of more than twenty)
  The end point of this secondary outcome considers a negative linear distribution for the correlation between PaO2/FiO2 and LUSS corrected by the presence of pleural effusions and pleural effusions' size.

CONTACTS AND LOCATIONS:
Overall Officials: Eleonore Vasseur, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (2):
- Belgium (2):
  - Centres Hospitaliers de Jolimont, Haine-Saint-Paul, Hainaut
  - Cliniques universitaires saint luc, Brussels

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Volpicelli G, Mussa A, Garofalo G, Cardinale L, Casoli G, Perotto F, Fava C, Frascisco M. Bedside lung ultrasound in the assessment of alveolar-interstitial syndrome. Am J Emerg Med. 2006 Oct;24(6):689-96. doi: 10.1016/j.ajem.2006.02.013. PMID 16984837
- [Background] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Lichtenstein D, Meziere G, Biderman P, Gepner A, Barre O. The comet-tail artifact. An ultrasound sign of alveolar-interstitial syndrome. Am J Respir Crit Care Med. 1997 Nov;156(5):1640-6. doi: 10.1164/ajrccm.156.5.96-07096. PMID 9372688
- [Background] Mojoli F, Bouhemad B, Mongodi S, Lichtenstein D. Lung Ultrasound for Critically Ill Patients. Am J Respir Crit Care Med. 2019 Mar 15;199(6):701-714. doi: 10.1164/rccm.201802-0236CI. PMID 30372119
- [Background] Zieleskiewicz L, Cornesse A, Hammad E, Haddam M, Brun C, Vigne C, Meyssignac B, Remacle A, Chaumoitre K, Antonini F, Martin C, Leone M. Implementation of lung ultrasound in polyvalent intensive care unit: Impact on irradiation and medical cost. Anaesth Crit Care Pain Med. 2015 Feb;34(1):41-4. doi: 10.1016/j.accpm.2015.01.002. Epub 2015 Mar 5. PMID 25829314
- [Background] Brogi E, Bignami E, Sidoti A, Shawar M, Gargani L, Vetrugno L, Volpicelli G, Forfori F. Could the use of bedside lung ultrasound reduce the number of chest x-rays in the intensive care unit? Cardiovasc Ultrasound. 2017 Sep 13;15(1):23. doi: 10.1186/s12947-017-0113-8. PMID 28903756
- [Background] Lichtenstein D, Goldstein I, Mourgeon E, Cluzel P, Grenier P, Rouby JJ. Comparative diagnostic performances of auscultation, chest radiography, and lung ultrasonography in acute respiratory distress syndrome. Anesthesiology. 2004 Jan;100(1):9-15. doi: 10.1097/00000542-200401000-00006. PMID 14695718
- [Background] Agricola E, Bove T, Oppizzi M, Marino G, Zangrillo A, Margonato A, Picano E. "Ultrasound comet-tail images": a marker of pulmonary edema: a comparative study with wedge pressure and extravascular lung water. Chest. 2005 May;127(5):1690-5. doi: 10.1378/chest.127.5.1690. PMID 15888847
- [Background] Soldati G, Copetti R, Sher S. Sonographic interstitial syndrome: the sound of lung water. J Ultrasound Med. 2009 Feb;28(2):163-74. doi: 10.7863/jum.2009.28.2.163. PMID 19168766
- [Background] Jambrik Z, Monti S, Coppola V, Agricola E, Mottola G, Miniati M, Picano E. Usefulness of ultrasound lung comets as a nonradiologic sign of extravascular lung water. Am J Cardiol. 2004 May 15;93(10):1265-70. doi: 10.1016/j.amjcard.2004.02.012. PMID 15135701
- [Background] Ziskin MC, Thickman DI, Goldenberg NJ, Lapayowker MS, Becker JM. The comet tail artifact. J Ultrasound Med. 1982 Jan-Feb;1(1):1-7. doi: 10.7863/jum.1982.1.1.1. PMID 6152918
- [Background] Yue Lee FC, Jenssen C, Dietrich CF. A common misunderstanding in lung ultrasound: the comet tail artefact. Med Ultrason. 2018 Aug 30;20(3):379-384. doi: 10.11152/mu-1573. PMID 30167593
- [Background] Minana G, Nunez J, Banuls P, Sanchis J, Nunez E, Robles R, Mascarell B, Palau P, Chorro FJ, Llacer A. Prognostic implications of arterial blood gases in acute decompensated heart failure. Eur J Intern Med. 2011 Oct;22(5):489-94. doi: 10.1016/j.ejim.2011.01.014. Epub 2011 Feb 25. PMID 21925058
- [Background] Gupta B, Jain G, Chandrakar S, Gupta N, Agarwal A. Arterial Blood Gas as a Predictor of Mortality in COVID Pneumonia Patients Initiated on Noninvasive Mechanical Ventilation: A Retrospective Analysis. Indian J Crit Care Med. 2021 Aug;25(8):866-871. doi: 10.5005/jp-journals-10071-23917. PMID 34733025
- [Background] Fan E, Brodie D, Slutsky AS. Acute Respiratory Distress Syndrome: Advances in Diagnosis and Treatment. JAMA. 2018 Feb 20;319(7):698-710. doi: 10.1001/jama.2017.21907. PMID 29466596
- [Background] Via G, Lichtenstein D, Mojoli F, Rodi G, Neri L, Storti E, Klersy C, Iotti G, Braschi A. Whole lung lavage: a unique model for ultrasound assessment of lung aeration changes. Intensive Care Med. 2010 Jun;36(6):999-1007. doi: 10.1007/s00134-010-1834-4. Epub 2010 Mar 11. PMID 20221746
- [Background] Zhao Z, Jiang L, Xi X, Jiang Q, Zhu B, Wang M, Xing J, Zhang D. Prognostic value of extravascular lung water assessed with lung ultrasound score by chest sonography in patients with acute respiratory distress syndrome. BMC Pulm Med. 2015 Aug 23;15:98. doi: 10.1186/s12890-015-0091-2. PMID 26298866
- [Background] Bouhemad B, Liu ZH, Arbelot C, Zhang M, Ferarri F, Le-Guen M, Girard M, Lu Q, Rouby JJ. Ultrasound assessment of antibiotic-induced pulmonary reaeration in ventilator-associated pneumonia. Crit Care Med. 2010 Jan;38(1):84-92. doi: 10.1097/CCM.0b013e3181b08cdb. PMID 19633538
- [Background] Bouhemad B, Brisson H, Le-Guen M, Arbelot C, Lu Q, Rouby JJ. Bedside ultrasound assessment of positive end-expiratory pressure-induced lung recruitment. Am J Respir Crit Care Med. 2011 Feb 1;183(3):341-7. doi: 10.1164/rccm.201003-0369OC. Epub 2010 Sep 17. PMID 20851923
- [Background] Soummer A, Perbet S, Brisson H, Arbelot C, Constantin JM, Lu Q, Rouby JJ; Lung Ultrasound Study Group. Ultrasound assessment of lung aeration loss during a successful weaning trial predicts postextubation distress*. Crit Care Med. 2012 Jul;40(7):2064-72. doi: 10.1097/CCM.0b013e31824e68ae. PMID 22584759
- [Background] Pisani L, Vercesi V, van Tongeren PSI, Lagrand WK, Leopold SJ, Huson MAM, Henwood PC, Walden A, Smit MR, Riviello ED, Pelosi P, Dondorp AM, Schultz MJ; Lung Ultrasound Consortium. The diagnostic accuracy for ARDS of global versus regional lung ultrasound scores - a post hoc analysis of an observational study in invasively ventilated ICU patients. Intensive Care Med Exp. 2019 Jul 25;7(Suppl 1):44. doi: 10.1186/s40635-019-0241-6. PMID 31346914
- [Background] Song G, Qiao W, Wang X, Yu X. Association of Lung Ultrasound Score with Mortality and Severity of COVID-19: A Meta-Analysis and Trial Sequential Analysis. Int J Infect Dis. 2021 Jul;108:603-609. doi: 10.1016/j.ijid.2021.06.026. Epub 2021 Jun 17. PMID 34146693
- [Background] Peach RJ, Day WA, Ellingsen PJ, McGiven AR. Ultrastructural localization of Tamm-Horsfall protein in human kidney using immunogold electron microscopy. Histochem J. 1988 Mar;20(3):156-64. doi: 10.1007/BF01746679. PMID 3410739
- [Background] Todur P; Souvik Chaudhuri FNB Critical Care; Vedaghosh Amara FNB Critical Care; Srikant N, Prakash P. Correlation of Oxygenation and Radiographic Assessment of Lung Edema (RALE) Score to Lung Ultrasound Score (LUS) in Acute Respiratory Distress Syndrome (ARDS) Patients in the Intensive Care Unit. Can J Respir Ther. 2021 May 19;57:53-59. doi: 10.29390/cjrt-2020-063. eCollection 2021. PMID 34041358
- [Background] Li L, Yao Y, Liu S. The Value of Pulmonary Bedside Ultrasound System in the Evaluation of Severity and Prognosis of Acute Lung Injury. Comput Math Methods Med. 2022 Jan 27;2022:6471437. doi: 10.1155/2022/6471437. eCollection 2022. PMID 35126630
- [Background] Vasseur E, Moureau G, Fasseaux A, Peyskens L, Gendebien F, Thys F, Dupriez F. Correlation between hypoxaemia and lung ultrasound score in patients presenting to an emergency department with interstitial syndrome: a prospective physiological study. Crit Care Resusc. 2023 Oct 18;24(3):233-241. doi: 10.51893/2022.3.OA2. eCollection 2022 Sep 5. PMID 38046212
- [Background] Lambden S, Laterre PF, Levy MM, Francois B. The SOFA score-development, utility and challenges of accurate assessment in clinical trials. Crit Care. 2019 Nov 27;23(1):374. doi: 10.1186/s13054-019-2663-7. PMID 31775846
- [Background] Li L, Yang Q, Li L, Guan J, Liu Z, Han J, Chao Y, Wang Z, Yu X. [The value of lung ultrasound score on evaluating clinical severity and prognosis in patients with acute respiratory distress syndrome]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2015 Jul;27(7):579-84. doi: 10.3760/cma.j.issn.2095-4352.2015.07.008. Chinese. PMID 26138420
- [Background] Brogi E, Gargani L, Bignami E, Barbariol F, Marra A, Forfori F, Vetrugno L. Thoracic ultrasound for pleural effusion in the intensive care unit: a narrative review from diagnosis to treatment. Crit Care. 2017 Dec 28;21(1):325. doi: 10.1186/s13054-017-1897-5. PMID 29282107
- [Background] Vignon P, Chastagner C, Berkane V, Chardac E, Francois B, Normand S, Bonnivard M, Clavel M, Pichon N, Preux PM, Maubon A, Gastinne H. Quantitative assessment of pleural effusion in critically ill patients by means of ultrasonography. Crit Care Med. 2005 Aug;33(8):1757-63. doi: 10.1097/01.ccm.0000171532.02639.08. PMID 16096453
- [Background] Roch A, Bojan M, Michelet P, Romain F, Bregeon F, Papazian L, Auffray JP. Usefulness of ultrasonography in predicting pleural effusions > 500 mL in patients receiving mechanical ventilation. Chest. 2005 Jan;127(1):224-32. doi: 10.1378/chest.127.1.224. PMID 15653988
- [Background] Balik M, Plasil P, Waldauf P, Pazout J, Fric M, Otahal M, Pachl J. Ultrasound estimation of volume of pleural fluid in mechanically ventilated patients. Intensive Care Med. 2006 Feb;32(2):318. doi: 10.1007/s00134-005-0024-2. Epub 2006 Jan 24. PMID 16432674
- [Background] Remerand F, Dellamonica J, Mao Z, Ferrari F, Bouhemad B, Jianxin Y, Arbelot C, Lu Q, Ichai C, Rouby JJ. Multiplane ultrasound approach to quantify pleural effusion at the bedside. Intensive Care Med. 2010 Apr;36(4):656-64. doi: 10.1007/s00134-010-1769-9. Epub 2010 Feb 6. PMID 20140421